CLINICAL TRIAL: NCT01370538
Title: A Phase III Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Trial of 14 Day Treatment With Esomeprazole 20 mg Once Daily in Subjects With Frequent Heartburn
Brief Title: Efficacy of Esomeprazole in Patients With Frequent Heartburn
Acronym: NEXT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D961RC00002
Record Dates: First submitted 2011-06-01; First posted 2011-06-10 (Estimated); Results first posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-03

CONDITIONS: Heartburn
Keywords: Heartburn
MeSH Terms: conditions — Heartburn | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Esomeprazole 20 mg (Experimental)
  Interventions: Drug: Esomeprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — Nexium 20 mg administered as 22.3 mg of esomeprasole magnesium hydrate, capsule, oral dose

SUMMARY:
This study will investigate the efficacy of esomeprazole 20 mg once a day in the treatment of frequent heartburn

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant ,non-lactating females 18 years or older
* Experience heartburn at least 2 days a week
* Having heartburn that has responded to heartburn medication
* Must discontinue any current heartburn medications

Exclusion Criteria:

* Having a history of erosive esophagitis verified by endoscopy
* Having a history of GERD which was diagnosed by a physician
* Inability to take study medication or complete the study and all study procedures
* Subjects that have required more than one 14-day course of PPI treatment within the past 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tore Lind, MD, Study Director — AstraZeneca
Locations (10):
- United States (10):
  - Research site, Mobile, Alabama
  - Research site, San Francisco, California
  - Research site, Westlake Village, California
  - Research site, Lexington, Kentucky
  - Research site, Rochester, New York
  - Research site, Dakota Dunes, South Dakota
  - Research site, Nashville, Tennessee
  - Research site, Austin, Texas
  - Research site, San Angelo, Texas
  - Research site, West Jordan, Utah

REFERENCES:
- [Derived] Peura D, Le Moigne A, Wassel H, Pollack C. Analysis of the symptom response to esomeprazole 20 mg over days 1-4 of a 14-day course of treatment for frequent heartburn: results of two randomised controlled trials. BMJ Open Gastroenterol. 2019 Jun 21;6(1):e000278. doi: 10.1136/bmjgast-2019-000278. eCollection 2019. PMID 31297231
- [Derived] Peura DA, Le Moigne A, Wassel H, Pollack C. Sustained efficacy following resolution of frequent heartburn with an over-the-counter regimen of esomeprazole 20 mg or placebo for 14 days: two randomized trials. BMC Gastroenterol. 2018 May 22;18(1):69. doi: 10.1186/s12876-018-0790-2. PMID 29788903
- [Derived] Peura D, Le Moigne A, Pollack C, Nagy P, Lind T. A 14-day regimen of esomeprazole 20 mg/day for frequent heartburn: durability of effects, symptomatic rebound, and treatment satisfaction. Postgrad Med. 2016 Aug;128(6):577-83. doi: 10.1080/00325481.2016.1203236. Epub 2016 Jul 4. PMID 27331882
- [Derived] Peura DA, Traxler B, Kocun C, Lind T. Esomeprazole treatment of frequent heartburn: two randomized, double-blind, placebo-controlled trials. Postgrad Med. 2014 Jul;126(4):33-41. doi: 10.3810/pgm.2014.07.2781. PMID 25141241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From total of 526 screened subjects, 341 subjects were randomised. From 341 subjects 170 and 171 were allocated to Esomeprazole and Placebo respectively.
Groups:
- Esomeprazole: Esomeprazole magnesium trihydrate 22.3 mg
- Placebo: Placebo for Esomeprazole
Period: Overall Study
Arm/Group | Esomeprazole | Placebo
Started | 170 | 171
Patients Who Received Treatment | 165 | 161
Patients Who Completed Treatment | 151 | 152
Completed | 151 | 152
Not Completed | 19 | 19
Not completed — Voluntary Discontinuation by Subject | 3 | 2
Not completed — Eligibility criteria not fulfilled | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 8 | 5
Not completed — Development of study specific withdrawal | 1 | 1
Not completed — Lost to follow up | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Placebo | Total
Number analyzed (Participants) | 170 | 171 | 341
Age Continuous [Mean (Standard Deviation); unit: Years]
  All | 41.6 (14.0) | 42.8 (13.2) | 42.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 87 | 178
  Male | 79 | 84 | 163
Race/Ethnicity, Customized [Number; unit: Participants]
  WHITE | 111 | 120 | 231
  BLACK OR AFRICAN AMERICAN | 52 | 50 | 102
  NATIVE HAWAIIAN/PACIFIC ISLANDER | 1 | 0 | 1
  AMERICAN INDIAN/ALASKA NATIVE | 3 | 0 | 3
  OTHER | 3 | 1 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  HISPANIC OR LATINO | 24 | 25 | 49
  NOT HISPANIC OR LATINO | 55 | 46 | 101
  NOT REPORTED | 91 | 100 | 191

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heartburn Free 24 Hour Days During 14 Days of Randomized Treatment
Time Frame: From randomisation to day 14
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Percentage of heartburn free days
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 162 | 158
Percentage of heartburn free days | 46.79 (33.32) | 30.93 (28.86)

2. Secondary Outcome: Number of Subjects Reporting Heartburn 2 Days or Less During the 14 Days Randomized Treatment Period
Description: Treatment period is considered to be both weeks 1 and 2 between V3 and V4.
Time Frame: From randomisation to the day 14
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 162 | 158
Participants | 27 | 2

3. Secondary Outcome: Comparison of Number of Subjects With 0, 1, 2, 3 or 4 Days With no Heartburn Over Days 1 to 4 Between Esomeprazole 20 mg and Placebo
Description: The first 4 consecutive days subjects were on randomized treatment, between V3 and V4.
Time Frame: From randomisation to day 14
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 162 | 158
Participants
  Zero days | 55 | 77
  One day | 32 | 34
  Two days | 22 | 29
  Three days | 37 | 16
  Four days | 16 | 2

4. Secondary Outcome: Number of Subjects With Heartburn 1 Day or Less During the Final Week, Second Week, First Week of Treatment
Description: There were three separate 7 day time periods during the treatment period; The first week (days 1-7), the second week (days 8-14), and the last 7 consecutive days (last day subject reported and the prior 6). For a given subject, the second week and last 7 consecutive days are the same if the subject has recorded measurements for the entire 14 day treatment period. However, for subjects reporting anything less than 14 days the two will not be identical. For all three 7 day time periods, days when a subject did not call in (i.e., missing values) were imputed as a day with heartburn.
Time Frame: From randomisation to day 14
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 162 | 158
Participants
  Last 7 consecutive days | 40 | 17
  Second 7 calendar days | 38 | 13
  First 7 calendar days | 32 | 7

5. Primary Outcome: Percentage of Heartburn Free 24 Hour Days During 14 Days of Randomized Treatment
Time Frame: From randomisation to day 14
Population: Per-protocol analysis set
Measure: Mean (Standard Deviation); unit: Percentage of heartburn free days
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 142 | 140
Percentage of heartburn free days | 47.82 (33.23) | 28.83 (31.22)

ADVERSE EVENTS:
Description: Full analysis set (FAS) population was analyzed.
Arm/Group | Esomeprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/158
Other Adverse Events (participants affected / at risk) | 18/162 | 15/158
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole (N=162) | Placebo (N=158)
Nausea (Gastrointestinal disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Pain (General disorders) | 0 | 3
Pyrexia (General disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2
Blood glucose decreased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 1 | 2
Haemoglobin decreased (Investigations) | 2 | 1
Hepatic enzyme increased (Investigations) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Headache (Nervous system disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days